CLINICAL TRIAL: NCT07007260
Title: Effect of Niacinamide Supplementation in Primary Open-angle Glaucoma
Brief Title: Effect of Niacinamide Supplementation in Glaucoma
Acronym: NiSPoG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Responsible Party: Principal Investigator, Adina Turcu-Stiolica, Professor, University of Medicine and Pharmacy Craiova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NiSPoG
Record Dates: First submitted 2025-01-13; First posted 2025-06-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Primary Open-Angle Glaucoma (POAG)
Keywords: visual field progression; quality of life
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Primary Open-angle Glaucoma (Experimental): Patients aged 18 years or older with confirmed diagnosis of Primary Open angle Glaucoma (POAG) - following a complete ophthalmological examination (ocular tonometry, slit lamp ocular examination, visual field and Optical coherence tomography).
  Interventions: Dietary Supplement: niacinamide supplementation

INTERVENTIONS:
Dietary Supplement: niacinamide supplementation — Patients will take niacinamide supplementation (500mg) every day for 1 year

SUMMARY:
Niacinamide is a chemical derivative of niacin, also known as vitamin B3. Through its complex role in the energetic metabolism, it has been evaluated and proven useful in several neurodegenerative disorders, such as Alzheimer's disease. Its effect in glaucoma, an optic nerve disorder related to a high intraocular pressure, is not well defined, and requires more research.

The investigators aim to assess the physiological effects of niacinamide on specific markers (e.g., visual field parameters, retinal nerve fibre layer thickness, electrophysiological markers such as the latency of the P2 wave on Flash visually evoked potentials) and on the quality of life in primary glaucoma patients.

DETAILED DESCRIPTION:
100 subjects with primary open-angle glaucoma will be enrolled from two centres (CMI profesor doctor Liliana Mary Voinea Bucharest Eye Centre and SC Optispecs Med SRL TgJiu Eye Clinic).

Participant Selection P1. Inclusion criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Patients aged 18 years or older;
* Confirmed diagnosis of Primary Open angle Glaucoma (POAG) - following a complete ophthalmological examination (ocular tonometry, slit lamp ocular examination, visual field and Optical coherence tomography);
* Subject has provided signed and dated written informed consent before admission to the study.
* Subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.
* Participants need to have visual acuity of Snellen ≥ 6/12 (0.5) or better.
* Have performed at least two reliable VFs (SITA-Fast 24-2), with <33% fixation losses and <15% false positives
* Those taking NAM already will undergo a 1-month washout period before commencing the study.

P2. Exclusion criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Participants must not be pregnant or breastfeeding women;
* Investigator considers the subject unfit for the study as a result of medical history, physical examination, or screening tests;
* VF damage worse than -10dB in the best eye and -16dB in the worse eye or a paracentral spot with -10dB or less in any eye),
* IOP >35mmHg in any eye or a mean IOP of 30mmHg or higher (two measurements), •inability to perform VFs,
* those unwilling to abstain from NAM supplements,
* allergic to niacinamide/niacin,
* diagnosed with cancer in the last 5 years (except treated basal or squamous cell carcinoma),
* a history of liver disease or stomach ulcers,
* disease that prevents long-term follow-up,
* neurologic or other non-glaucomatous conditions apart from cataract that may affect the VF
* Patient is diagnosed with primary angle closure glaucoma;
* Patient is diagnosed with secondary glaucoma (e.g. posttraumatic, postinflammatory, steroid induced, pseudoexfoliative, pigmentary, etc.);
* Patient is diagnosed with very advanced glaucoma (foveal fixation threatened or absent and, thus, unreliable perimetry);
* Patient is diagnosed with other significant ocular pathologies (advanced cataract, pathologic myopia, corneal ectasias or dystrophies, sever amblyopia, vitreoretinal disease, active ocular inflammation, significant sequelae of ocular inflammation);
* Unreliable ophthalmological investigations and non-compliance with examinations (e.g. high percentage of false negative and false positive errors when examining the visual field).

Participants will:

* Take NAM every day for 1 year
* Visit the clinic at 3, 6, and 12 months for check-ups and tests

Outcome Measures M1. Ophthalmological parameters

* Visual field parameters:

  * Mean deviation (MD)
  * Pattern standard deviation (PSD)
* Optical coherence tomography parameters: peripapillary retinal nerve fiber layer thickness (pRNFL);
* Visually evoked potential parameter: latence of P2 wave when using a flash stimulus.

M2. Quality of life measurement

➔ Glaucoma Quality of Life-15 questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Confirmed diagnosis of Primary Open angle Glaucoma (POAG) - following a complete ophthalmological examination (ocular tonometry, slit lamp ocular examination, visual field and Optical coherence tomography); Subject has provided signed and dated written informed consent before admission to the study.
* Subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.
* Participants need to have visual acuity of Snellen ≥ 6/12 (0.5) or better.
* Have performed at least two reliable VFs (SITA-Fast 24-2), with <33% fixation losses and <15% false positives
* Those taking NAM already will undergo a 1-month washout period before commencing the study.

Exclusion Criteria:

* Participants must not be pregnant or breastfeeding women;
* Investigator considers the subject unfit for the study as a result of medical history, physical examination, or screening tests;

  •● VF damage worse than -10dB in the best eye and -16dB in the worse eye or a paracentral spot with -10dB or less in any eye),
* OP >35mmHg in any eye or a mean IOP of 30mmHg or higher (two measurements), •inability to perform VFs,
* those unwilling to abstain from NAM supplements,
* allergic to NAM/niacin,
* diagnosed with cancer in the last 5 years (except treated basal or squamous cell carcinoma),
* a history of liver disease or stomach ulcers,
* disease that prevents long-term follow-up, neurologic or other non-glaucomatous conditions apart from cataract that may affect the VF
* Patient is diagnosed with primary angle closure glaucoma;
* Patient is diagnosed with secondary glaucoma (e.g. posttraumatic, post inflammatory, steroid induced, pseudo exfoliative, pigmentary, etc.);
* Patient is diagnosed with very advanced glaucoma (foveal fixation threatened or absent and, thus, unreliable perimetry);
* Participants who are currently on NAM will be asked to stop taking the tablets for a month prior to screening visit.
* Patient is diagnosed with other significant ocular pathologies (advanced cataract, pathologic myopia, corneal ectasias or dystrophies, sever amblyopia, vitreoretinal disease, active ocular inflammation, significant sequelae of ocular inflammation);
* Unreliable ophthalmological investigations and non-compliance with examinations (e.g. high percentage of false negative and false positive errors when examining the visual field).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
logMAR | 3, 6 and 12 months from the baseline
  Ophthalmological parameters
  ➔ Visual field parameters: logMAR

SECONDARY OUTCOMES:
QoL | 3, 6 and 12 months from the baseline
  Glaucoma Quality of Life-15 questionnaire responses (Subtirelu, M.S., Nicola, C.A.; Turcu-Stiolica, M.; Turcu-Stiolica, A. Translation and Cultural Adaptation of the Glaucoma Quality of Life-15 Questionnaire to the Romanian Population. Value in Health 2023, Volume 26, Issue 6, S318-S319)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy of Craiova, Craiova, Dolj, Romania

REFERENCES:
- [Derived] Nicola CA, Marinescu MC, Firan AM, Tartea G, Naidin MS, Ciuluvica RC, Dimulescu MD, Voicu NM, Mihailescu CM, Meca AD, Bogdan M, Turcu-Stiolica A. Changes in Quality of Life Among Glaucoma Patients Following Six Months of Niacinamide Supplementation. Nutrients. 2025 Aug 27;17(17):2775. doi: 10.3390/nu17172775. PMID 40944166